CLINICAL TRIAL: NCT05679141
Title: Clinical Correlation Between Self-collected and Physician-collected HPV Screening Kits
Status: Completed | Type: Observational
Sponsor: Switch Health Solutions Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HPV102022
Record Dates: First submitted 2022-12-07; First posted 2023-01-10 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: HPV Infection; Cervical Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to validate the of the Evalyn®Brush via self-collection to the standard clinician-collected technique using the BD SurePath™ collection vial and Rovers CombiBrush for detection of Human Papillomavirus (HPV). This study will validate the sensitivity and specificity of the Evalyn Brush with the future goal of making this testing approach available for self-collection in the future.

DETAILED DESCRIPTION:
Cervical cancer is one of the most common female cancers in the world. It has been reported that approximately 1300 Canadians are diagnosed with cervical cancer each year. HPV is a common sexually transmitted DNA virus comprised of more than 100 genotypes. Ninety seven percent (97%) of cervical cancer is attributed to 12 strains of HPV and 70% of cervical cancer cases across the world are attributed to 2 specific strains of the virus (HPV 16 and 18).

The current screening practice in Canada is to use cytology-based testing (Pap testing) for primary screening to detect signs of abnormal cervical cells. However, this is dependent on access and willingness to see a trained clinician for a pelvic exam and cervical cell collection.

HPV testing aims to detect the presence of HPV DNA or RNA. It requires 2 components: adequate sample collection and PCR based testing. Most HPV screening programs are dependent on clinician collected samples, however, self-collected vaginal samples may improve access to testing and thus, overall impact of screening programs.

Many studies have been completed to assess the viability of self-collected samples for HPV testing as compared to clinical collected samples. In a randomized, controlled trial (RCT), women who were attending a clinical for a routine pap test and pelvic exam were included in the study to assess the effectiveness of vaginal self-sampling. The swab self-collection method was found to be non-inferior compared to the clinical specimen. The tampon method of collection, however, was not equivalent.

Results from an Italian pilot study showed self-collected samples demonstrated adequate cellularity (cells stability and health) with the devices tested. HPV testing of self-collected vaginal samples using semi-automated vs automated systems shows good concordance with clinician-collected cervical sample.

CADTH published a Horizon Scan in 2021. (Canada's Drug and Health Technology Agency, 2021) Table 1 is a summary of the evidence they reviewed. There were no safety issues reported for these HPV self-collection devices.

Many studies have assessed the impact of self-collected sampling on increased access and willingness to test in high-risk, underprivileged, or otherwise reluctant populations. One such by Desai et all found that the implementation of self-collect vaginal testing in a Nigerian population, increased screening rates to over 100 women per clinic day, making way for early treatment planning as needed. Reques et al.noted the potential for this approach in an under-served population of France.

Expanding sample collection opportunities beyond existing clinical environments is anticipated to improve access and frequency of HPV screening. Accordingly, cases may be identified earlier in the prognosis, leading to earlier intervention and better health outcomes.

Switch Health has performed a review to identify and evaluate potential collection devices and laboratory protocols for HPV. The Rovers Evalyn®Brush has been selected as the preferred candidate for initial pilot and validation. A 'dry' media was preferred over other liquid media as the use of dry samples eliminates issues related to liquid medium such as spillage, skin irritation, or accidental consumption. Additionally, spillage of the liquid media, by the user or in the lab, can affect the analytical volume for analysis and may impact the accuracy of results. Dry samples can be mailed directly to the lab without any other major considerations (such as Transportation of Dangerous Goods) and at a lower cost, as compared to an equivalent liquid sample.

The Rovers Evalyn® Brush has been designed for self-collection of vaginal samples and may be as accurate as clinician-collected cervical samples. This study will validate the accuracy of the Evalyn® Brush (clinician-collected) with the purpose of making this testing approach available for self-collection in the future.

Expanding sample collection opportunities beyond existing clinical environments to self-collected samples is anticipated to increase testing frequency due to convenience and access. Accordingly, cases may be identified earlier in the prognosis leading to earlier intervention and better health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant visiting the study site for a potential OB/GYN purpose
* Participant >= 21 years of age
* Participant has a cervix

Exclusion Criteria:

* Currently menstruating
* Currently pregnant or within 3 months following pregnancy
* Utilized vaginal products within past 48 hrs.
* Experiencing any of following symptoms:

Pain in lower abdomen Fever Unusual or heavy vaginal discharge Pain / bleeding when having intercourse Painful or frequent urination

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population are individuals with a cervix who wish to participate in routine screening for HPV and associated risk for cervical cancers.
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Clinical Correlation - Positives | Through study completion, an average of 12 weeks
  Samples collected via self-collection correlate >95% to those clinician-collected
Clinical Correlation - Negatives | Through study completion, an average of 12 weeks
  Samples collected via self-collection correlate >95% to those clinician-collected

CONTACTS AND LOCATIONS:
Overall Officials: Karam Ramotar, PHD, Principal Investigator — Bio-Test Laboratory
Locations (1):
- Ottawa Medical Group, Ottawa, Ontario, Canada